CLINICAL TRIAL: NCT00571610
Title: A Single-Center, Open-Label, Single-Arm Pilot Study of the Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty Implantable Device Used to Reduce Mitral Valve Regurgitation.
Brief Title: Montreal Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty Device
Acronym: PTOLEMY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viacor (Industry)
Responsible Party: Katharine M Stohlman, Viacor, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-020P
Record Dates: First submitted 2007-11-30; First posted 2007-12-12 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Heart Failure; Mitral Regurgitation
Keywords: Heart Failure; Mitral Regurgitation
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patient is screened for study and given baseline assessments. Patient receives a diagnostic PTMA assessment and if responsive, receives a PTMA implant.
  Interventions: Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant

INTERVENTIONS:
Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant — Percutaneous access from right or left subclavian vein, diagnostic assessment, then placement of the PTMA implant in the coronary sinus, great cardiac vein.

SUMMARY:
Reduction in mitral regurgitation due to safe placement of a PTMA device in the coronary sinus.

ELIGIBILITY:
Inclusion Criteria:

* Functional MR 2+ - 4+ with left ventricular enlargement
* Symptomatic heart failure
* 20% - 50% LVEF

Exclusion Criteria:

* mitral regurgitation of organic origins
* recent cardiac interventions
* severe comorbidities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
percent of patients who remain free from device-related major adverse events (death, myocardial infarction, tamponade, emergent cardiac surgery | 30 days

SECONDARY OUTCOMES:
percent of implanted patients who maintain a sustained 1 grade reduction in MR and reduction of mitral annulus anterior posterior dimension | 30 days
percent of implanted patients who exhibit improvement of clinical symptoms as one of the following: decrease in NYHA class, improvement of Minnesota QOL survey, increase exercise capacity 6 minute walk or improvement in VO2 max | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Luc Bilodeau, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Dubreuil O, Basmadjian A, Ducharme A, Thibault B, Crepeau J, Lam JY, Bilodeau L. Percutaneous mitral valve annuloplasty for ischemic mitral regurgitation: first in man experience with a temporary implant. Catheter Cardiovasc Interv. 2007 Jun 1;69(7):1053-61. doi: 10.1002/ccd.21186. PMID 17525965